CLINICAL TRIAL: NCT03073551
Title: The Impact of Activity Promoting Video Games on Glycemic Control in Gestational Diabetes Mellitus
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 10-188
Record Dates: First submitted 2017-02-03; First posted 2017-03-08 (Actual); Last update posted 2020-04-29 (Actual); Status verified 2020-04

CONDITIONS: Gestational Diabetes Mellitus
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Intervention Model Description: The control group will receive diabetes treatment and education as per standard of care.
  The intervention group will receive diabetes treatment and education as per standard of care, and will also be given a Wii game console to bring home.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Participants in this group will receive diabetic care and education as per the standard of care. They will also be given a pedometer and will be instructed to record their number of steps at the end of each day
- Wii Group (Active Comparator): Participants in this group will receive diabetic care and education as per the standard of care. They will also be given a Wii console and game to take home. Participants will be instructed on how to set up and use the Wii. These participants will also be given a pedometer and will be instructed to record their number of steps at the end of each day.
  Interventions: Other: Wii Group

INTERVENTIONS:
Other: Wii Group — Participants in the Wii group will be given a Wii console and video game to take home. The console includes a Wii balance board and remote controller. The Wii Fit game allows participants to choose different types of exercise such as yoga, aerobics, balance training, and more. Participant movements are shown on screen as they move with the balance board and remote control.
  Arms: Wii Group

SUMMARY:
Gestational diabetes mellitus (GDM) affects up to 3-5% of all pregnancies. When diagnosed with GDM, women undergo nutritional counseling, blood sugars monitoring and are encouraged to exercise regularly. Women who do not meet therapeutic targets may need to add insulin injections. Activity promoting video games are an attractive possibility for improvement of exercise compliance. The objective of this study is to determine whether providing women recently diagnosed with GDM with a Nintendo Wii™ activity promoting gaming platform will increase activity levels, improve glycemic control of sugar levels and decrease the need for supplementary insulin treatment.

DETAILED DESCRIPTION:
As part of the standard of care, all pregnant women are screened with a 50 gram glucose challenge test between 24-28 weeks gestation. Women are diagnosed with GDM when they have two abnormal values on the 75 gram oral glucose tolerance test. Once a diagnosis of GDM has been made women are referred to the diabetes in pregnancy clinic within 1-2 weeks. All women initially undergo a group session with a clinical nutritionist and a registered nurse specializing in diabetic care. During this session women receive basic information regarding gestational diabetes, instruction regarding dietary management of GDM and standard recommendations regarding physical activity. Women also routinely receive a glucometer for self monitoring of glucose levels and are instructed regarding its use. One week after this group session an intake session with an endocrinologist and Maternal-Fetal Medicine specialist occurs and glycemic control is reviewed. Follow up visits are scheduled every 1-4 weeks depending on adequacy of glycemic control. Decisions regarding adequacy of dietary management and need for insulin therapy are made by the endocrinologist at each subsequent visit.

For the purpose of our study, patients will be approached after this group teaching session. Eligible patients who have consented to participate in the study will undergo randomization into two groups:

1. Control - routine GDM care as mentioned above.
2. Intervention - This group will undergo all aspects of routine GDM care but will also receive a Nintendo Wii gaming console + Wii Fit activity platform. The games provided include "Wii sport" and Wii Fit Plus". Each participant will receive a 30-60 minute guided information session to ensure that she is able to install the console at home and to set up her personal login information. At this session an overview of the available Wii activities will be presented. Each participant will receive a telephone number to call in case technical difficulties are encountered at home. At 36 weeks of gestation, the Wii hardware and programs will be returned to the investigators. Participants will be instructed to note the following warning signs for termination of the exercise session; vaginal bleeding, dyspnea before exertion, dizziness, headache, chest pain, muscle weakness, calf pain or swelling, preterm labor, decreased fetal movement, and amniotic fluid leakage.

As mentioned, all participants in the study will be encouraged to be physically active. In order to independently calculate and compare the overall level of physical activity in both groups all participating women will receive a pedometer (StepsCount Digi-Walker SW700) and will be instructed to wear it daily during waking hours.

ELIGIBILITY:
Inclusion Criteria:

* Women diagnosed with gestational diabetes and a singleton pregnancy at 24-36 weeks of gestation.

Exclusion Criteria:

* Multiple gestation
* Pre-gestational diabetes
* Unable to provide informed consent
* Any contraindication to performing physical activity in pregnancy (e.g. increased risk of preterm delivery)
* Has and regularly uses a Nintendo Wii console
* Presence of co-morbidities including: Hypertension (systolic pressure > 160 mmHg and/or diastolic pressure > 100 mmHg), alcohol abuse (i.e. 2 glasses alcohol or more per day); drug abuse, use of the medication that affects insulin secretion or insulin sensitivity (antiviral, corticosteroids, antihypertensive drugs, all concomitant medication will be discussed); serious pulmonary (COPD, exercise induced asthma), cardiac, hepatic or renal (serum creatinine > 150 μmol/l) impairment; malignant disease; serious mental or physical impairment (limiting the ability to understand or implement the study protocol).

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Participants must be pregnant women
Enrollment: 150 (Actual)
Dates: Start 2010-07-27 (Actual); Primary Completion 2022-08-01 (Estimated); Study Completion 2022-08-01 (Estimated)

PRIMARY OUTCOMES:
Glucose levels | Measured from study intake date until 36 weeks gestation
  Mean fasting and post-prandial glucose levels

SECONDARY OUTCOMES:
Insulin therapy | Measured from study intake date until 36 weeks gestation
  Need for insulin therapy to control insulin levels
Activity level | Measured from study intake date until 36 weeks gestation
  Level of daily physical activity performed
Maternal weight gain | Weight gained during pregnancy, measured from start of pregnancy (1 week gestation) to end of pregnancy (up to 40 weeks gestation).
  Measured as the amount of weight gained from time of conception to time of delivery

CONTACTS AND LOCATIONS:
Overall Officials: Howard Berger, MD, Principal Investigator — Unity Health Toronto

IPD SHARING:
Plan to Share IPD: No